CLINICAL TRIAL: NCT00878891
Title: Real Time Continuous Glucose Monitoring With Glucoday® as an Assistant for Intensive Insulin Therapy in Diabetic Cardiothoracic Surgery Patients: a Randomized Study Comparing Blood Glucose Measurements Alone or Associated to Continue Glucose Monitoring
Brief Title: Real-time Continuous Glucose Monitoring in Diabetic Cardiothoracic Surgery Patients
Acronym: MARGE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Menarini Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CHUBX 2007/01
Record Dates: First submitted 2009-04-08; First posted 2009-04-09 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2015-07

CONDITIONS: Diabetes
Keywords: Microdialysis; realtime; glucose sensor; coronary artery bypass
MeSH Terms: conditions — Diabetes Mellitus | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1. Conventional glucose monitoring (Active Comparator): Discontinuous glucose monitoring - GlucoDay Device with Continue record blinded
  Interventions: Device: Continuous glucose monitoring for immediate correction of abnormal glycemia
- 2. Conventional glucose monitoring + Glucoday (Experimental): Continuous glucose monitoring - GlucoDay device with Continue record displayed
  Interventions: Device: Continuous glucose monitoring for immediate correction of abnormal glycemia

INTERVENTIONS:
Device: Continuous glucose monitoring for immediate correction of abnormal glycemia — Prevention of hyper and hypo glycemia

SUMMARY:
An increased risk of adverse outcome is noted for diabetic patients admitted in surgery intensive care units (ICU). Tight glycemic control with intensive insulin therapy dramatically reduces in-hospital mortality and adverse outcome. Devices recording continuously interstitial glucose monitoring (CGM) may be an aid in patients of ICU in whom normoglycemia become a target.

The mini-invasive device (Glucoday®) should provide real-time glucose concentrations in order to quickly adjust insulin infusion rates. The objective of MARGE study is to compare percent of time in normoglycemia based on conventional monitoring (discontinuous glucose monitoring) and Glucoday to conventional monitoring alone. The MARGE study is a multicenter (2 centers), randomized, single blind trial.

Several studies have shown that hyperglycemia is associated with poor outcomes in hospitalized patients. Postoperative glucose levels are a significant predictor of infection rates after cardiac surgery and death rate. Based on these observational studies, a randomized controlled intervention trial in surgical ICU patients demonstrated that intensive insulin therapy reduced the overall in-hospital mortality by 34 % and stream infection by 46 %. Using continuous glycemic monitoring (CGM) it has been shown that intensive insulin therapy based on discontinuous glucose monitoring revealed that normoglycemia is achieved only 22 % of time. The researchers' aim is to determine if real time CGM with a new generation mini invasive device, Glucoday® S, would allow quickly adjusting insulin infusions rates according to interstitial glucose levels and decreasing both hyperglycemic and hypoglycemic excursions. This study will further investigate whether application of real time CGM to titrate insulin therapy to target glycemia in a tight range (80-110 mg/dl) can improve diabetic patient outcome after coronary artery bypass grafting (CABG).

DETAILED DESCRIPTION:
Diabetes is a major and independent risk factor of coronary disease. Coronary artery bypass graft (CABG) significantly improves the patients' prognostic. However postoperative hyperglycemia is a morbidity and mortality factor.

Tight glycemic control with intensive insulin therapy dramatically reduces in-hospital mortality and adverse outcome but with a significant risk of hypoglycaemia. Intensive discontinuous blood glucose control may be insufficient to adapt insulin doses to reach ambitious glycemia targets in safety. Therefore new tools are needed for glucose monitoring in diabetic patients admitted in surgery intensive care units (ICU). The mini-invasive continuous interstitial glucose monitoring device Glucoday® (Menarini Diagnostics) has been recently developed and allows to access continuous interstitial glucose monitoring with real time record display.

The primary outcome measure: is the Comparison of post CABG glycemia in diabetic patients treated by intensive insulin therapy either by conventional monitoring (discontinuous capillary glucose monitoring), or by conventional monitoring and CGM using GlucoDay®. The principal criterion of glycemic control is the percent of time spent in normoglycemia (0.8 - 1.10 g/L).

The secondary outcome measures: are 1: Comparison of percent of post CABG time in hyperglycemia (>1.8 g/l) and hypoglycemia (<0.5 g/l) in the two randomization groups. 2: Comparison of clinical outcomes incidence during 30 days after CABG: death rate, cardiovascular events (acute coronary syndromes, heart failure, arrhythmia) stream infections, neurologic events. 3: Comparison of performance and accuracy between CGM with Glucoday® and conventional capillary blood glucose monitoring in the setting of CABG and surgical ICU. 4: Comparison of duration of stay in ICU and in the surgical care unit. 5: Description of device and care tolerance by collection of all adverse events due to the device during the hospitalization

Study design: It's an efficacy multi-center randomized clinical trial with parallel assignment. The principal analysis will be performed on all patients and if the difference is clinically significant, it will be performed on sub-groups.

Inclusion criteria are Patients aged from 20 to 80 years, patients admitted for CABG ,patients with Known type 1 and type 2 diabetes, patients with Type 2 diabetes discovered during surgical or anaesthetic pre-operative consultation (plasmatic glycemia > 1.26 g/l) needing only dietary guidelines, Patients affiliated to the French Social Security and informed consent signed

Exclusion criteria are patients with other types of cardiac surgery than CABG, Patients admitted in emergency, Pregnancy or breastfeeding for woman, Patients included in an other clinical trial with an exclusion period still running, Patients under safeguard of justice

Study procedures:

* Arm 1. conventional glucose monitoring (discontinuous glucose monitoring)
* Arm 2. conventional glucose monitoring + GlucoDay® (continuous glycemic monitoring)

Primary efficacy end-points: percent of time spent in normoglycemia (0.80-1.10 g/l) between the end of the surgical intervention and 48 hours after the first device calibration (performed after the intervention)

Principal secondary efficacy end-points: 1: percent of time in hyperglycemia (> 1.8 g/l) and in hypoglycaemia (<0.5g/l) between time of intervention and 48 hours after the first device calibration. 2: composite criterion evaluated one month after inclusion: death or cardiovascular event events (acute coronary syndromes, heart failure, arrhythmia) stream infections, neurologic events. 3: agreement between CGM with Glucoday® and conventional capillary blood glucose monitoring using coupled data recorded at the same time except couples of data corresponding to calibration time (T0, T24H). 4: duration of stay in hospital for the two randomization groups. 5: device and care tolerance by collection of all adverse events due to the device during the hospitalization.

The enrollment: is 154 patients, 77 in each group

Flow chart:

At the screening visit, patients are informed about the study, eligibility criteria are verified and standard laboratory analyses are performed. At the inclusion visit (one day before surgical intervention), eligibility criteria are verified, the informed consent is signed, standard laboratory analyses, clinical exam and randomization are performed. At day 0, The CABG is performed and the patients are transferred to ICU where Glucoday® is installed. At day 2 (48 hours) Glucoday® is removed. At day 7, a clinical exam is performed. Between CABG and day 30 all events are collected.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged from 20 to 80 years
* Admitted for CABG
* Type 2 diabetes
* Type 1 diabetes
* Type 2 diabetes discovered during surgical or anaesthetic pre-operative consultation (plasmatic glycemia > 1.26 g/l) needing only dietary guidelines
* Informed consent signed
* Patients affiliated to the french social security

Exclusion Criteria:

* Other types of cardiac surgery than CABG
* Patients admitted in emergency
* Pregnancy or breastfeeding
* Patients included in an other clinical trial with an exclusion period still running
* Patients under safeguard of justice

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2009-04; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Percent of time in normoglycemia (0.8 - 1.10 g/L) | Between the hour of the end of the intervention (CABG) and T48 hours after the first calibration of the Glucoday or while battery last

SECONDARY OUTCOMES:
Percent of post CABG time in hyperglycemia (>1.8 g/l) and hypoglycemia (<0.5 g/l) | Between the hour of the end of the intervention (CABG) and T48 hours after the first calibration of the Glucoday or while battery last
Clinical outcomes incidence : death rate, cardiovascular events (acute coronary syndromes, heart failure, arrhythmia) stream infections, neurologic events | during 30 days after CABG
Agreement between CGM with Glucoday and conventional capillary blood glucose monitoring in the setting of CABG and surgical ICU | During 48 hours
During of stay in ICU and in tyhe surgical care unit | During the hospitalisation
Adverse events due to the device | During the hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Bogdan CATARGI, MD PHD, Principal Investigator — University Hospital Bordeaux, France
Locations (1):
- Service d'endocrinologie-Diabétologie - Hôpital Haut-Lévêque - CHU de Bordeaux, Pessac, France

REFERENCES:
- [Background] Calafiore AM, Di Mauro M, Di Giammarco G, Contini M, Vitolla G, Iaco AL, Canosa C, D'Alessandro S. Effect of diabetes on early and late survival after isolated first coronary bypass surgery in multivessel disease. J Thorac Cardiovasc Surg. 2003 Jan;125(1):144-54. doi: 10.1067/mtc.2003.73. PMID 12538998
- [Background] Capes SE, Hunt D, Malmberg K, Gerstein HC. Stress hyperglycaemia and increased risk of death after myocardial infarction in patients with and without diabetes: a systematic overview. Lancet. 2000 Mar 4;355(9206):773-8. doi: 10.1016/S0140-6736(99)08415-9. PMID 10711923
- [Background] Furnary AP, Gao G, Grunkemeier GL, Wu Y, Zerr KJ, Bookin SO, Floten HS, Starr A. Continuous insulin infusion reduces mortality in patients with diabetes undergoing coronary artery bypass grafting. J Thorac Cardiovasc Surg. 2003 May;125(5):1007-21. doi: 10.1067/mtc.2003.181. PMID 12771873
- [Background] Furnary AP, Zerr KJ, Grunkemeier GL, Starr A. Continuous intravenous insulin infusion reduces the incidence of deep sternal wound infection in diabetic patients after cardiac surgical procedures. Ann Thorac Surg. 1999 Feb;67(2):352-60; discussion 360-2. doi: 10.1016/s0003-4975(99)00014-4. PMID 10197653
- [Background] Koschinsky T, Heinemann L. Sensors for glucose monitoring: technical and clinical aspects. Diabetes Metab Res Rev. 2001 Mar-Apr;17(2):113-23. doi: 10.1002/dmrr.188. PMID 11307176
- [Background] Malmberg K. Prospective randomised study of intensive insulin treatment on long term survival after acute myocardial infarction in patients with diabetes mellitus. DIGAMI (Diabetes Mellitus, Insulin Glucose Infusion in Acute Myocardial Infarction) Study Group. BMJ. 1997 May 24;314(7093):1512-5. doi: 10.1136/bmj.314.7093.1512. PMID 9169397
- [Background] Malmberg K, Norhammar A, Wedel H, Ryden L. Glycometabolic state at admission: important risk marker of mortality in conventionally treated patients with diabetes mellitus and acute myocardial infarction: long-term results from the Diabetes and Insulin-Glucose Infusion in Acute Myocardial Infarction (DIGAMI) study. Circulation. 1999 May 25;99(20):2626-32. doi: 10.1161/01.cir.99.20.2626. PMID 10338454
- [Background] Malmberg K, Ryden L, Wedel H, Birkeland K, Bootsma A, Dickstein K, Efendic S, Fisher M, Hamsten A, Herlitz J, Hildebrandt P, MacLeod K, Laakso M, Torp-Pedersen C, Waldenstrom A; DIGAMI 2 Investigators. Intense metabolic control by means of insulin in patients with diabetes mellitus and acute myocardial infarction (DIGAMI 2): effects on mortality and morbidity. Eur Heart J. 2005 Apr;26(7):650-61. doi: 10.1093/eurheartj/ehi199. Epub 2005 Feb 23. PMID 15728645
- [Background] Maran A, Crepaldi C, Tiengo A, Grassi G, Vitali E, Pagano G, Bistoni S, Calabrese G, Santeusanio F, Leonetti F, Ribaudo M, Di Mario U, Annuzzi G, Genovese S, Riccardi G, Previti M, Cucinotta D, Giorgino F, Bellomo A, Giorgino R, Poscia A, Varalli M. Continuous subcutaneous glucose monitoring in diabetic patients: a multicenter analysis. Diabetes Care. 2002 Feb;25(2):347-52. doi: 10.2337/diacare.25.2.347. PMID 11815508
- [Background] McAlister FA, Man J, Bistritz L, Amad H, Tandon P. Diabetes and coronary artery bypass surgery: an examination of perioperative glycemic control and outcomes. Diabetes Care. 2003 May;26(5):1518-24. doi: 10.2337/diacare.26.5.1518. PMID 12716815
- [Background] Van den Berghe G. How does blood glucose control with insulin save lives in intensive care? J Clin Invest. 2004 Nov;114(9):1187-95. doi: 10.1172/JCI23506. PMID 15520847
- [Background] van den Berghe G, Wouters P, Weekers F, Verwaest C, Bruyninckx F, Schetz M, Vlasselaers D, Ferdinande P, Lauwers P, Bouillon R. Intensive insulin therapy in critically ill patients. N Engl J Med. 2001 Nov 8;345(19):1359-67. doi: 10.1056/NEJMoa011300. PMID 11794168